CLINICAL TRIAL: NCT00002623
Title: RANDOMIZED TRIAL OF SURGERY VERSUS RADIOTHERAPY IN PATIENTS WITH STAGE IIIa NON-SMALL CELL LUNG CANCER AFTER A RESPONSE TO INDUCTION-CHEMOTHERAPY
Brief Title: Chemotherapy Followed by Surgery or Radiation Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-08941; EORTC-08941
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed during surgery. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether chemotherapy followed by surgery with or without radiation therapy is more effective than chemotherapy followed by radiation therapy alone in treating non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy followed by surgery with or without radiation therapy to that of chemotherapy followed by radiation therapy alone in treating patients who have stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with stage IIIA non-small cell lung cancer treated with surgery with or without radiotherapy versus radiotherapy alone after achieving a response to a neoadjuvant chemotherapy regimen containing cisplatin or carboplatin.
* Compare the progression-free survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, response to induction chemotherapy (complete vs partial vs minor), and histological subtype (squamous vs nonsquamous).

All patients receive 3 courses of induction combination chemotherapy comprising cisplatin or carboplatin in the absence of disease progression or unacceptable toxicity. Patients with complete or partial response (or minor response if disease has become resectable) are randomized to 1 of 2 treatment arms.

* Arm I: Within 6 weeks of randomization, patients undergo radical lobectomy or pneumonectomy plus dissection of the hilar and mediastinal lymph nodes.

Patients with positive resection margins of at least 1 cm and/or positive mediastinal nodes undergo radiotherapy 5 days a week for 5.5 weeks.

Patients with postresection subclinical/microscopic disease with negative tumor margins undergo radiotherapy 5 days a week for 4-4.5 weeks.

* Arm II: Within 6 weeks of randomization, patients undergo primary radiotherapy. Patients with subclinical/microscopic disease with negative tumor margins undergo radiotherapy 5 days a week for 4-4.5 weeks.

Patients with gross tumor volume and tumor margins at least 1 cm undergo radiotherapy 5 days a week for 6 weeks.

Patients are followed every 3 months for 2 years and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 640 patients will be accrued for this study within 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven primary unresectable non-small cell lung cancer (NSCLC) by mediastinoscopy, mediastinotomy, thoracotomy, video-assisted thoracic surgery, or needle biopsy

  * Stage IIIA (N2) disease by chest CT scan
  * Any histologic subtype allowed
* At least 1 unidimensionally or bidimensionally measurable target lesion on chest CT scan
* No N3 or metastatic disease by physical exam, CT scan of thorax, bone scan, and CT scan or ultrasound of liver and adrenals
* No pre-existing pleural or pericardial effusion
* No symptomatic CNS involvement

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No superior vena cava syndrome

Pulmonary:

* No diffuse interstitial pulmonary fibrosis

Other:

* No prior melanoma, breast cancer, or hypernephroma
* No other primary malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix
* No grade 2 or greater pre-existing motor or sensory neurotoxicity
* No active uncontrolled infection requiring IV antibiotics
* Must be physically and mentally fit for study therapy
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for NSCLC

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for NSCLC

Surgery:

* No prior surgery for NSCLC

Other:

* No other prior therapy for NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 1994-12; Primary Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ted A.W. Splinter, MD, Study Chair — University Medical Center Rotterdam at Erasmus Medical Center
Locations (30):
- Belgium (8):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Hopital de Jolimont, Haine-Saint-Paul
  - U.Z. Gasthuisberg, Leuven
  - CHR - Clinique Saint Joseph - Hopital de Warqueguies, Mons
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
  - Stedelijk Ziekenhuis, Roesclare
- Academisch Ziekenhuis Utrecht, Vandœuvre-lès-Nancy, France
- Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova), Italy
- Netherlands (17):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Ziekenhuis St Jansdal, Harderwijk
  - Atrium Medical Centre, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Leiden University Medical Center, Leiden
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - University Medical Center Nijmegen, Nijmegen
  - Saint Franciscus Ziekenhuis, Roosendaal
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Erasmus Medical Center, Rotterdam
  - Twee Steden Ziekenhuis Vestiging Tilburg, Tilburg
  - Diakonessenhuis Utrecht, Utrecht
  - Sophia Ziekehuis, Zwolle
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester, England
  - Royal Marsden Hospital, Sutton, England
  - Royal Victoria Hospital, Belfast, Northern Ireland

REFERENCES:
- [Background] Van Meerbeeck JP, De Pauw R, Tournoy K. What is the optimal treatment of stage IIIA-N2 non-small-cell lung cancer after EORTC 08941? Expert Rev Anticancer Ther. 2008 Feb;8(2):199-206. doi: 10.1586/14737140.8.2.199. PMID 18279061
- [Result] van Meerbeeck JP, Kramer GW, Van Schil PE, Legrand C, Smit EF, Schramel F, Tjan-Heijnen VC, Biesma B, Debruyne C, van Zandwijk N, Splinter TA, Giaccone G; European Organisation for Research and Treatment of Cancer-Lung Cancer Group. Randomized controlled trial of resection versus radiotherapy after induction chemotherapy in stage IIIA-N2 non-small-cell lung cancer. J Natl Cancer Inst. 2007 Mar 21;99(6):442-50. doi: 10.1093/jnci/djk093. PMID 17374834
- [Result] Kramer GW, Legrand CL, van Schil P, Uitterhoeve L, Smit EF, Schramel F, Biesma B, Tjan-Heijnen V, van Zandwijk N, Splinter T, Giaccone G, van Meerbeeck JP; EORTC-Lung Cancer Group. Quality assurance of thoracic radiotherapy in EORTC 08941: a randomised trial of surgery versus thoracic radiotherapy in patients with stage IIIA non-small-cell lung cancer (NSCLC) after response to induction chemotherapy. Eur J Cancer. 2006 Jul;42(10):1391-8. doi: 10.1016/j.ejca.2006.01.052. PMID 16785054
- [Result] Van Meerbeeck JP, Kramer GW, Legrand C, et al.: Does downstaging in patients (pts) with IIIA-N2 non-small cell lung cancer (NSCLC) and a response to induction chemotherapy (ICT) influence outcome with surgery (S) or radiotherapy (RT)? An exploratory analysis of EORTC 08941. [Abstract] J Clin Oncol 24 (Suppl 18): A-7047, 375s, 2006.
- [Result] Van Meerbeeck JP, Kramer G, Van Schil PE, et al.: A randomized trial of radical surgery (S) versus thoracic radiotherapy (TRT) in patients (pts) with stage IIIA-N2 non-small cell lung cancer (NSCLC) after response to induction chemotherapy (ICT) (EORTC 08941). [Abstract] J Clin Oncol 23 (Suppl 16): A-LBA7015, 624s, 2005.
- [Result] Van Schil P, Van Meerbeeck J, Kramer G, Splinter T, Legrand C, Giaccone G, Manegold C, van Zandwijk N. Morbidity and mortality in the surgery arm of EORTC 08941 trial. Eur Respir J. 2005 Aug;26(2):192-7. doi: 10.1183/09031936.05.00127204. PMID 16055865
- [Result] van Meerbeeck JP, Kramer GWPM, van Schil PEY, et al.: Induction chemotherapy (CT) in stage IIIA-N2 non-small cell lung cancer (NSCLC):an analysis of different regimens used in EORTC 08941. [Abstract] Lung Cancer 41 (Suppl 2): A-O-273, S79, 2003.
- [Result] van Schil PE, van Meerbeeck JP, Kramer G, et al.: Surgery after induction chemotherapy: morbidity and mortality in the first 100 patients of the surgery arm of EORTC 08941 trial. [Abstract] Lung Cancer 41 (Suppl 2): A-O-147, S45, 2003.
- [Result] Splinter TA, van Schil PE, Kramer GW, van Meerbeeck J, Gregor A, Rocmans P, Kirkpatrick A. Randomized trial of surgery versus radiotherapy in patients with stage IIIA (N2) non small-cell lung cancer after a response to induction chemotherapy. EORTC 08941. Clin Lung Cancer. 2000 Aug;2(1):69-72; discussion 73. doi: 10.3816/clc.2000.n.020. PMID 14731343